CLINICAL TRIAL: NCT04858932
Title: Novel Digital Endpoints in Geriatric Anorexia
Brief Title: Geriatric Anorexia Study
Acronym: GAS
Status: Completed | Type: Observational
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Other Study IDs: H-40837
Record Dates: First submitted 2021-04-14; First posted 2021-04-26 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Healthy
Keywords: Healthy; Wearable Devices; Geriatric Anorexia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Fried Frailty Phenotype 0: Those who are considered Robust under the Fried Frailty Criteria. Sensor technology and digital measures will be used to evaluate movement, metabolism, body weight composition, glucose levels, and nutritional scale in healthy adults.
  Interventions: Device: Continuous Glucose Monitor; Device: Wrist Actigraphy Device; Device: Food Weight Scale; Device: Smart Body Weight Scale
- Fried Frailty Phenotype 1-2: Those who are considered Intermediate/Pre-frail under the Fried Frailty Criteria. Sensor technology and digital measures will be used to evaluate movement, metabolism, body weight composition, glucose levels, and nutritional scale in healthy adults.
  Interventions: Device: Continuous Glucose Monitor; Device: Wrist Actigraphy Device; Device: Food Weight Scale; Device: Smart Body Weight Scale
- Fried Frailty Phenotype 3+: Those who are considered Frail under the Fried Frailty Criteria. Sensor technology and digital measures will be used to evaluate movement, metabolism, body weight composition, glucose levels, and nutritional scale in healthy adults.
  Interventions: Device: Continuous Glucose Monitor; Device: Wrist Actigraphy Device; Device: Food Weight Scale; Device: Smart Body Weight Scale

INTERVENTIONS:
Device: Continuous Glucose Monitor — a handheld reader and a wearable sensor placed on the back of the arm used to obtain glucose measurements
  Other Names: Freestyle Libre
Device: Wrist Actigraphy Device — a watch like wearable sensor
  Other Names: Geneactiv Watch
Device: Food Weight Scale — a scale to measure food weight
  Other Names: Renpho
Device: Smart Body Weight Scale — a full body composition scale that provides fat and muscle mass, water retention, bone mass, and weight trends
  Other Names: Renpho

SUMMARY:
Reduction in appetite and/or food intake among older individuals is referred to as anorexia of aging (AOA, also known as Geriatric Anorexia). AOA is linked with myriad comorbidities associated with aging, contributes significantly to adverse health consequences in old age, and has been used as a predictor of morbidity and mortality. The overall aim of this study is to assess the feasibility and burden of the proposed in-laboratory and out-of-laboratory assessments to study Geriatric Anorexia. This will be accomplished with the use of questionnaires as well as devices that evaluate movement, metabolism, body weight composition, glucose levels, and nutritional scale.

DETAILED DESCRIPTION:
This is a study to evaluate movement, metabolism, body weight composition, glucose levels, and nutritional scale in healthy adults. Subjects, age 65 to 85 years will be recruited.

The proposed study will consist of an initial (in-clinic) intake visit on Day 1 where the subject will be screened and enrolled in the study after signing an informed consent document, followed by an at-home phase where the subject will wear a watch like device on one wrist. After training, the subject will return for their Day 8 in-clinic visit, where the subject will repeat some intake assessments and activities, as well as some additional standing and walking activities. The subject will then be asked to perform at-home activities and assessments with the use of a smart phone, digital food scale, smart body weight scale, and continuous glucose monitor, while continuing to wear the watch-like device and a movement measurement device around their waist (Days 8-21). A final in-clinic visit will take place on Day 21 for final assessments and device collection. A +/- 4 days will be allocated for the scheduling of all visits to accommodate subject's schedules and commitments. All in-laboratory activities will take place in the Laboratory for Human Neurobiology while in-home activities will be completed in the subject's home. The study procedures will be identical for all subjects for the three groups.

ELIGIBILITY:
Inclusion Criteria:

[separated into the three groups based on the Fried Criteria: 0, 1-2, 3 or above]

* Male or female participants aged 65 - 85 years.
* No clinically significant health problems other than well controlled chronic conditions (e.g., allergies and dermatitis)
* No recent hospitalizations/acute events in last 12 months.
* No active or recent (within 12 months) cancer diagnosis except skin cancer (limited to only non-complicated Squamous Cell Carcinoma (SCC)/Basal Cell Carcinoma (BCC)).
* Body mass index (BMI) < 30 kg/m2
* Able to understand and cooperate with study procedures and able to read, understand and provide informed consent. Evidence of a personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study
* Participants should not have any food aversion which could influence their food selection if standardized meals are used as part of the protocol.
* Native English speakers or demonstrated fluency in English as determined by the Investigator.
* Wide Range Achievement Test (WRAT-4) Word Reading Subtest equivalent to 8th grade reading level or greater.
* Normal or corrected-to-normal vision

Exclusion Criteria:

* Treatment with an investigational drug within 30 days of enrollment
* A moderate to severe alcohol use disorder diagnosis within 6 months of the screening as disclosed by the subject
* Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Boston University/Boston Medical Center directly involved in the conduct of the study
* Inability to comply with study requirements.
* Has any clinically significant medical disorder, condition, disease or clinically significant finding at screening that precludes subject's participation in study activities including any self-reported diagnosis of eating disorders.
* Participants with electronic implant devices, such as pacemaker.
* Non-English Reader as measured by the WRAT-4.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Assess the feasibility, usability, and compliance of wearing a GENEActiv watch in a geriatric population both in-clinic and remotely at-home. | 21 days +/- 4 days
  One GENEActiv watch will be used on one wrist and one around the waist at a sampling rate of 50 Hz to measure movement in the x, y, and z direction across the study period.
Assess the feasibility, usability, and compliance of food consumption tracking in a geriatric population both in-clinic and remotely at-home. | 21 days +/- 4 days
  A food scale will be used to track food consumed in grams (g) throughout the study. The total number of meals consumed per day and across study period.
Assess the feasibility, usability, and compliance of body weight composition measurements in a geriatric population both in-clinic and remotely at-home. | 21 days +/- 4 days
  A body weight composition scale will be used to completion of daily weight measurement and track body weight in kilograms (kg) throughout the study.
Assess the correlation of a GENEActiv watch with frailty phenotype in elderly participants. | 21 days +/- 4 days
  One GENEActiv watch will be used on one wrist and one around the waist at a sampling rate of 50 Hz to measure movement in the x, y, and z direction. This data will be compared to frailty phenotype per the Fried Frailty Scale and continuous glucose measurements.
Assess the correlation of food consumption with frailty phenotype in elderly participants. | 21 days +/-4 days
  A food scale will be used to track food consumed in grams (g) throughout the study. This data will be compared to frailty phenotype per the Fried Frailty Scale.
Assess the correlation of the body weight composition scale with frailty phenotype in elderly participants. | 21 days +/-4 days
  A body weight composition scale will be used to track body weight in kilograms (kg) throughout the study. This data will be compared to frailty phenotype per the Fried Frailty Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Thomas, PhD, MBA, Principal Investigator — Principal Investigator, Boston University, Department of Anatomy & Neurobiology
Locations (1):
- Evans Biomedical Research Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided